CLINICAL TRIAL: NCT00314171
Title: A Study of a Glaucoma Therapy to Treat Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-05-10
Record Dates: First submitted 2006-04-10; First posted 2006-04-13 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2012-03

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: open-angle glaucoma; ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Timolol; Ophthalmic Solutions; Suspensions; dorzolamide; Solutions; dorzolamide-timolol combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brinzolamide + Timolol (Experimental)
  Interventions: Drug: Brinzolamide 10 mg/ml + Timolol 5 mg/ml eye drops, suspension
- Dorzolamide + Timolol (Active Comparator)
  Interventions: Drug: Dorzolamide 20 mg/ml + Timolol 5 mg/ml eye drops, solution (COSOPT)

INTERVENTIONS:
Drug: Brinzolamide 10 mg/ml + Timolol 5 mg/ml eye drops, suspension — One drop in the study eye(s) twice daily for 12 months
  Arms: Brinzolamide + Timolol
Drug: Dorzolamide 20 mg/ml + Timolol 5 mg/ml eye drops, solution (COSOPT) — One drop in the study eye(s) twice daily for 12 months
  Other Names: COSOPT
  Arms: Dorzolamide + Timolol

SUMMARY:
The purpose of this study is to determine whether a glaucoma therapy is safe and effective in treating patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosis of open-angle glaucoma or ocular hypertension
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Under 18
* Pregnant
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2005-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Mean IOP

SECONDARY OUTCOMES:
Percent patients with IOP < 18 mmHg

REFERENCES:
- [Result] Manni G, Denis P, Chew P, Sharpe ED, Orengo-Nania S, Coote MA, Laganovska G, Volksone L, Zeyen T, Filatori I, James J, Aung T. The safety and efficacy of brinzolamide 1%/timolol 0.5% fixed combination versus dorzolamide 2%/timolol 0.5% in patients with open-angle glaucoma or ocular hypertension. J Glaucoma. 2009 Apr-May;18(4):293-300. doi: 10.1097/IJG.0b013e31818fb434. PMID 19365194